CLINICAL TRIAL: NCT00528203
Title: Comprehensive Sickle Cell Centers (CSCC) Collaborative Genotype-Phenotype Database and Sample Repository
Brief Title: Establishing a Repository of Blood and DNA Samples From People With Sickle Cell Disease (Comprehensive Sickle Cell Centers Collaborative Genotype-Phenotype Database and Sample Repository)
Acronym: Gen/Phen
Status: Terminated | Type: Observational
Why Stopped: Funds for study ended September 30, 2008.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Carolyn Hoppe, MD, Children's Hospital Oakland
Other Study IDs: 517; U54HL070587 (NIH)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-11

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Sickle Cell Anemia; DNA
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Lymphocytes, Whole blood, RBC hemolysate, DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited blood disease that can cause intense pain episodes. The purpose of this study is to collect, test, and archive blood and DNA samples from children and adults with SCD to study the role that genes play in SCD. Blood and DNA samples will be stored for use in future SCD studies.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder that is caused by an abnormal type of hemoglobin. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." The Comprehensive Sickle Cell Centers (CSCC) is a network of 10 centers that conduct research to improve health care and treatment options for people with SCD. The Collaborative Data Project (C-Data) is a CSCC study that is establishing a comprehensive database of children and adults with SCD who are receiving medical care at participating CSCC research centers. This study will initiate the development of a centralized laboratory that will collect, test, and archive blood and DNA samples from participants in the C-Data project for use in future SCD studies. The collection of blood and DNA samples will provide researchers with an important resource to better define the genetic diversity of SCD. In the future, genotype-phenotype correlation studies, population studies, and various other genetic studies may be conducted.

This study will enroll participants taking part in the C-Data project. For this study, participants will undergo a blood collection. The blood sample will then be sent to a lab to characterize the red blood cells and hemoglobin. DNA will be analyzed to identify genes that influence the severity of SCD. Blood and DNA will be stored for future genetic research in SCD and closely related disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the C-Data project

Exclusion Criteria:

* Unable to undergo blood collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and pediatric patients who are enrolled in the C-Data project are eligible for this study. (C-Data eligibility: All adult and pediatric patients who have been seen within the last 24 months in the hospital or clinical setting and are expected to return episodically or regularly for care at 1 of the CSCC are eligible for inclusion in the C-Data project.)
Sampling Method: Non-Probability Sample
Enrollment: 3640 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Hoppe, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (13):
- United States (13):
  - Children's Hospital Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital of Boston, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Medical Hospital of Dallas, Dallas, Texas
  - University of Texas Southwestern & Parkland, Dallas, Texas
  - University of Texas at Galveston, Galveston, Texas